CLINICAL TRIAL: NCT00392522
Title: 50% Nitrous Oxide and 50% Oxygen (MEOPA) Conscious Sedation Versus Placebo in Fiberoptic Bronchoscopy : Randomized, Double Blind, Placebo-Controlled Study
Brief Title: 50% Nitrous Oxide and 50% Oxygen (MEOPA) Conscious Sedation Versus Placebo in Fiberoptic Bronchoscopy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004.417
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2007-10

CONDITIONS: Fiberoptic Bronchoscopy
Keywords: Anxiety; Cough; Number of general anaesthesias (due to procedure failure); Patients satisfaction; Chest physician satisfaction
MeSH Terms: conditions — Anxiety Disorders; Cough | interventions — Nitrous Oxide; Oxygen; Meopa

INTERVENTIONS:
Drug: 50% Nitrous Oxide and 50% Oxygen (MEOPA)

SUMMARY:
Fiberoptic bronchoscopy may generate pain, anxiety or cough and dyspnea. It may then induce discomfort and then run down its yield. Systematic local anaesthesia does not always suffice and FOB may be conducted under general anaesthesia. Premixed nitrous oxide and oxygen (MEOPA) could be efficient to avoid general anesthesia risks and to reduce organizational costs. Nitrous oxide induces anaelgesia and anxiolysis when administered in oxygen at a 50% concentration.

MEOPA is being delivered in France for every short painful medical in-patients procedure since 2001. At a concentration of 50% in oxygen, and delivered through a facial mask, it produces a conscious sedation useful during endoscopy. MEOPA safety is due to its short term effect, which ends 5 minutes after cessation of inhalation. It therefore allows ambulatory medicine.

Two randomized double blind controlled studies were driven in fiberoptic bronchoscopy (Fauroux 2004, Atassi 2005) and showed its efficacy on pain control and sedation.

We will perform our Study to estimate MEOPA efficacy in term of pain control (Visual Analogic Scale (VAS)), anxiety control (COVI Scale), cough and number of general anaesthesias, comparing FOB under MEOPA and Oxygen (double blind, randomized, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 who should undergo a fiberoptic bronchoscopy (inpatient and outpatient)

Exclusion Criteria:

* Child under 18
* Pneumothorax
* ocular surgery in the previous 3 months,
* intracranial overpressure
* lucidity impairment
* emphysema bullae
* face trauma
* angina pectoris
* hemodynamic instability
* acute respiratory distress
* hypercapnia > 45 mm Hg
* pregnancy
* lidocaine allergia
* lack of approuval from the patient to perform the study will of the patient to undergo FOB with premixed nitrous oxide-oxygen

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2006-11

PRIMARY OUTCOMES:
Efficacy in term of pain control Visual Analogic Scale

SECONDARY OUTCOMES:
anxiety control (COVI Scale)
cough
number of general anaesthesias

CONTACTS AND LOCATIONS:
Overall Officials: Corinne DEPAGNE, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Corinne Depagne, Lyon, France